CLINICAL TRIAL: NCT00942864
Title: An Open-label, Nonrandomized, Phase IIIb, Single Dose Study to Evaluated the Changes in Optical Coherence Tomography (OCT) and Fluorescein Angiography (FA) After Intravitreal Injection of Lucentis® in Patients With Macular Edema Secondary to Retinal Vein Occlusion (RVO)
Brief Title: Effect of Intravitreal Ranibizumab Injection With Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Korea Ltd. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002AKR07
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab

INTERVENTIONS:
Drug: ranibizumab — ranibizumab 0.5mg (0.05ml volume), intravitreal injection first 3 injection every 4 weeks additional injection (optional) according to the judgement of doctor
  Other Names: Lucentis®

SUMMARY:
The purpose of this study is to evaluate the effects of intravitreal Lucentis® (Ranibizumab) and investigate the anatomical and functional improvement following this treatment in patients with macular edema due to retinal vein occlusion (RVO).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with macular edema due to RVO (confirmed by fundus photography, fluorescein angiography, OCT)
* Male and female aged from 18 to 70
* Baseline best-corrected visual acuity (BCVA) in the study eye was from 20/400 to 20/30 using ETDRS chart

Exclusion Criteria:

* Additional eye disease that could compromise VA
* Ocular inflammation
* Intraocular surgery ≤ 1 month before day 0
* Uncontrolled glaucoma
* Prior treatments with laser photocoagulation or other intervention for macular edema due to BRVO
* Patients aged under 18 or over 71
* Female patient in pregnancy or breast feeding
* Not suitable to regular follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The change in ETDRS visual acuity letter scores from baseline. The change in the 1-mm central retinal thickness as measured by OCT from baseline. | every 4 weeks (up to 52 weeks)

SECONDARY OUTCOMES:
The intraretinal structure changes in OCT. Progression of avascular area by FA. Number of additional treatments. Intraocular safety (endophthalmitis, uveitis, increase in intraocular pressure, etc). | every 4 weeks (up to 52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Young Yu, Principal Investigator — Dept. ophthalmology, Kyunghee medical center
Locations (1):
- Dept. of ophthalmology, Kyung Hee University Medical Center, Seoul, South Korea